CLINICAL TRIAL: NCT00978601
Title: Improved Recovery Using Multimodal Peri-operative Analgesia in Minimally Invasive Myomectomy.A Randomized Study.
Brief Title: Improved Recovery Using Multimodal Peri-operative Analgesia in Minimally Invasive Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iakentro Fertility Centre (Other)
Responsible Party: Panos Xiromeritis MD, Iakentro Advanced Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MULTI-LM-100
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Anesthesia; Myomectomy
Keywords: post-operative analgesia; early discharge,; fast recovery,; minimally invasive myomectomy,; laparoscopy,; laparoscopically assisted myomectomy; patient discharge; Anesthesia Recovery Period

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodal analgesic protocol group (Experimental): Women who received the multimodal analgesic protocol during minimally invasive myomectomy.
  Interventions: Procedure: Multimodal analgesic protocol during minimally invasive myomectomy
- No use of multimodal analgesic protocol group (No Intervention): Women who did not receive the multimodal analgesic protocol during minimally invasive myomectomy.
  Interventions: Procedure: Multimodal analgesic protocol during minimally invasive myomectomy

INTERVENTIONS:
Procedure: Multimodal analgesic protocol during minimally invasive myomectomy — Multimodal and preemptive analgesia using 8 mg of Dexamethasone iv,trocar ports infiltration with 5 mL of a local anesthetic, consisting of 0.26% ropivacaine HCL (7.5 mg/mL) and 0.74% of 0,9 % sodium chloride, before the skin incision. About 10 minutes before the surgery is completed, 4 mg Ondansetron iv and a mixture of 75 mg diclofenac and 600 mg of paracetamol intramuscularly (im) are administered.

SUMMARY:
The purpose of this study is to evaluate a multimodal analgesic protocol used in minimally invasive surgery for myomectomies (laparoscopic myomectomy (LM) and laparoscopically assisted myomectomy (LAM)).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic intramural and or subserous myomas
* ASA score 1-2
* Without contraindication to nonsteroidal anti-inflammatory agents
* Patients have to be able to understand and follow medical instructions
* They need to have satisfactory hygiene and accommodation conditions
* They have to live not more than 2 hours away from the department
* Easy telephone contact is required

Exclusion Criteria:

* Ovarian disease
* Previous medical treatment for ovarian suppression, pregnancy, abnormal Papanicolaou (Pap) test smear or hyperplasia (with or without atypia) in case of endometrial biopsy

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The main outcome measure is the Visual Analog Scale (VAS) score at 2 and 8 hours post surgery. | 2 and 8 hours post surgery.

SECONDARY OUTCOMES:
hours of the bowel peristalsis return, hours of hospitalization, and number of days for the fully recuperate activity are also measured. | hours to few days after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Iakentro Advanced Medical Center, Thessaloniki, Greece

REFERENCES:
- [Background] de Lapasse C, Rabischong B, Bolandard F, Canis M, Botchorischvili R, Jardon K, Mage G. Total laparoscopic hysterectomy and early discharge: satisfaction and feasibility study. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):20-5. doi: 10.1016/j.jmig.2007.08.608. PMID 18262139
- [Background] Prapas Y, Kalogiannidis I, Prapas N. Laparoscopy vs laparoscopically assisted myomectomy in the management of uterine myomas: a prospective study. Am J Obstet Gynecol. 2009 Feb;200(2):144.e1-6. doi: 10.1016/j.ajog.2008.08.063. Epub 2008 Nov 18. PMID 19019334
- [Background] Hoffman CP, Kennedy J, Borschel L, Burchette R, Kidd A. Laparoscopic hysterectomy: the Kaiser Permanente San Diego experience. J Minim Invasive Gynecol. 2005 Jan-Feb;12(1):16-24. doi: 10.1016/j.jmig.2004.12.022. PMID 15904592
- [Background] Kehlet H, Wilkinson RC, Fischer HB, Camu F; Prospect Working Group. PROSPECT: evidence-based, procedure-specific postoperative pain management. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):149-59. doi: 10.1016/j.bpa.2006.12.001. PMID 17489225
- [Derived] Xiromeritis P, Kalogiannidis I, Papadopoulos E, Prapas N, Prapas Y. Improved recovery using multimodal perioperative analgesia in minimally invasive myomectomy: a randomised study. Aust N Z J Obstet Gynaecol. 2011 Aug;51(4):301-6. doi: 10.1111/j.1479-828X.2011.01333.x. Epub 2011 Jul 5. PMID 21806591